CLINICAL TRIAL: NCT05632640
Title: Effectiveness of Weighted Blankets to Decrease Emergence Agitation, Sedation, and Vascular Complications in a Pediatric Cardiac Post Anesthesia Care Unit Following Cardiac Catheterization
Brief Title: Post Anesthesia Care Unit (PACU) Weighted Blanket Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Brian J Armstrong, Registered nurse and principal investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00215568
Record Dates: First submitted 2022-11-09; First posted 2022-11-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Catheterization; Electrophysiology Procedure; Pediatric Cardiology
Keywords: weighted blanket; post anesthesia care unit; recovery; agitation; pediatrics; Pediatric Cardiology; Emergence delirium
MeSH Terms: conditions — Psychomotor Agitation; Emergence Delirium | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of Care
- Weighted blanket (Experimental)
  Interventions: Device: Weighted blanket

INTERVENTIONS:
Other: Standard of Care — Following the participants procedure, standard of care will be given in the recovery area.
  Arms: Standard of Care
Device: Weighted blanket — Following the participants procedure once in the recovery area, the nursing staff will place a weighted blanket on the participants. Different weighted blanket sizes will be used based on participants weight.
  Arms: Weighted blanket

SUMMARY:
This study is being conducted to evaluate the safety and efficacy of weighted blankets to reduce agitation in patients in the post-procedural phase after cardiac catheterization and electrophysiology procedures in the post anesthesia care unit.

The study hypothesizes that compared to the traditional and current post-procedural strategy, weighted blanket use will reduce agitation and therefore lessen the need for additional sedation along with a reduction of post-procedure vascular complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac catheterization or electrophysiology procedure
* Post Procedure bedrest plan for greater than (>)2 hours
* Duration of recovery planned for 11th floor cardiac PACU

Exclusion Criteria:

* Patients less than (<) 40 pounds (18 kilogram (kg))
* Patients > 220 pounds (100 kg)
* Recovery anticipated to not be in our cardiac PACU
* Posttraumatic stress disorder
* Claustrophobia
* Uncontrolled seizure disorders
* Open heart surgery within 30 days
* Severe pulmonary hypertension
* Severe asthma
* Sleep apnea requiring continuous positive airway pressure (CPAP)
* Known diaphragm paresis
* Home vent/CPAP
* Restrictive lung disease (such as patients with scoliosis)
* Higher risk for upper respiratory airway occlusion (such as patients with Down Syndrome)
* Cast, brace or splint, fractures
* Degenerative muscular disorder (such as patients with cerebral palsy)
* Areas of impaired skin integrity
* Gastrostomy tube
* Percutaneous endoscopic gastrostomy
* Tracheostomy
* Chest tube(s)
* PACU procedures required (within 1 hour post arrival): post operative (post op) echocardiogram, post op Xray, post op electrocardiogram

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Average Richmond Agitation Sedation Scale (RASS) compared between the two groups | up to 60 minutes (after arrived to PACU)
  Richmond Agitation Sedation Score is a validated and standardized scoring system ranging from negative 5 (unarousable sedation) to 0 (awake and calm) to 4 (combative).

SECONDARY OUTCOMES:
Analgesia administered in the recovery area | up to 6 hours after arriving in the PACU
  Number of medications (Midazolam, Ketamine, Propofol, Dexmedetomidine, Lorazepam, etc.) required during the recovery period following the procedure.
Incidence of vascular complications in the recovery area | up to 6 hours after arriving in the PACU
  This will include participants that have episodes of re-bleeding and hematomas.
Safety measures assessed by vital sign parameters for absolute oxygen (O2 saturation) | up to 6 hours after arriving in the PACU
  Absolute oxygen (O2) saturation drop of 10 points or more from recovery area arrival baseline.
Safety measures assessed by vital sign parameters for respiration rate | up to 6 hours after arriving in the PACU
  Respiration rate decreased 20% or more from recovery arrival baseline.
Safety measures assessed by vital sign parameters for respiratory effort | up to 6 hours after arriving in the PACU
  Increased Respiratory Effort (retractions, labored, nasal flaring, etc.) as compared to recover area arrival baseline

CONTACTS AND LOCATIONS:
Overall Officials: Brian Armstrong, RN, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No